CLINICAL TRIAL: NCT03084341
Title: Effectiveness of Two Stretching Techniques on Healthy Volunteers With Shortened Hamstrings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Jorge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04/2016
Record Dates: First submitted 2016-11-07; First posted 2017-03-20 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Muscle Tone Abnormalities
Keywords: Elasticity; Electric Stimulation; Muscle Stretching Exercises
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NMEE Group (Active Comparator): Neuromuscular Electrical Elongation
  Interventions: Procedure: Neuromuscular Electrical Elongation
- PNF Group (Active Comparator): Proprioceptive Neuromuscular Facilitation stretching
  Interventions: Procedure: Proprioceptive Neuromuscular Facilitation
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Procedure: Neuromuscular Electrical Elongation — Electrotherapy equipment will be used, choosing an interferential current through bipolar application,with a frequency of 4 kHz and a frequency modulation amplitude of 100 Hz.
  Arms: NMEE Group
Procedure: Proprioceptive Neuromuscular Facilitation — Hold-relax technique that involves lengthening the muscle to the point of limitation, at which point the individual performs an isometric contraction for up to 10 s, followed by a passive movement of the limb into the new end-range.
  Arms: PNF Group

SUMMARY:
The main objective of this study is to compare the effect and the duration of the Neuromuscular Electrical Elongation (NMEE ) technique versus the PNF technique and versus a control group, on the extensibility of the hamstrings muscles.

Hypothesis:

NMEE of shortened hamstrings muscles in healthy subjects, compared with PNF and control group produces a significant increase in hamstrings extensibility.

DETAILED DESCRIPTION:
It is a double-blinded randomized clinical trial where subjects are healthy volunteers from the city of Zaragoza older than 18 years. All subjects will be injury free at the time of the study and must not have a history of knee or hip surgery. They must be physically active, but without engaging in competition-level sports, and must have flexibility deficits, as measured in the AKE test position and SLK test position (<60º AKE; < 80º SLK).

There will be an NMEE Group (Neuromuscular Electrical Elongation), an PNF Group (Proprioceptive Neuromuscular Facilitation) and a Control Group (No Invervention).

Intervention:

NMEE technique will be performed by stretching the muscle till resistance and applying a bipolar interferential current to produce an involuntary contraction of the muscle which will be maintained 3 seconds. After that, the subject will contract the antagonist muscle (quadriceps) actively until he feels resistance again . Then, intensity of the electrical current is increased again. This cycle will be repeated 4 times.

PNF technique will be performed by stretching the muscle till resistance is felt. Then the patient will have to make an isometric contraction of the muscle (against resistance) during 3 seconds. After that, the subject will contract the antagonist muscle (quadriceps) actively until he feels resistance again. This contract-stretch cycle will be repeated 4 times.

Control group: This group will not receive a training program.

In case of shortening, the assigned intervention will be performed until the values considered normal with a maximum of 8 stretching sessions (2 per week). Otherwise, if there is no shortening, the intervention will end at that moment.

Assessment:

To assess the effectiveness of these techniques several tests will be performed on the subjects.

For hamstrings extensibility:

* Active-Knee-Extension Test (AKE) results will bring information of the knee extension range of motion.
* Straight-Leg-Raise Test (SLR) results will bring information of the hip flexion range of motion.

For quadriceps extensibility:

* Goniometric measure of knee flexion.
* Distance from heel to gluteus using a tape measure.

Viscoelasticity properties of hamstrings and quadriceps muscles:

- Myotonometric measurement using a myotonometer to obtain frequency, decrement (elasticity) and stiffness.

For neural assessment:

- The Slump Test is a neural tension test used to detect altered neurodynamics or neural tissue sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers
* Older than 18 years
* Bilateral shortened hamstrings muscles with a knee extension under 60º (TEAR, Neto et al., 2015) and a ROM under 80º in the hip (straight leg raise test angle, Espejo-Antúnez et al., 2015)

Exclusion Criteria:

* Participation in a muscular stretching program during the study
* Previous history of surgical intervention in the hip, tight or knee
* Muscle-skeletal pain or injury in the low back or inferior limbs
* Abdominal o spine surgery within three month before the study beginning.

Exit Criteria:

* Patient´s petition
* Change in the regular physical activity level during the study period
* Appearance of an injury that would contraindicate the use of stretching techniques

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Active-knee-extension test (AKE) | Pre-intervention; Post-intervention (30 minutes after intervention); Follow up (4 week after last intervention)
  The AKE is performed using an experimental apparatus designed specifically for this investigation. It consists of a rectangular wooden frame that is attached to an examination table. The tested limb is flexed until the thigh touched the wooden frame, being at 90° with the table. The contralateral limb is fully extended and stabilized in neutral rotation by a second examiner. With the foot in neutral position and the knee flexed at 90°, a standard universal goniometer is placed over the lateral femoral condyle, with 1 arm aligned along the thigh in direction to the greater trochanter and the other arm aligned over the leg in the direction of the lateral malleolus.
  From this position, and without any prior warm-up subjects will be instructed to extend the knee until they felt a strong resistance, holding this final position for 2 to 3 seconds to allow the goniometric reading.
Change in Straight-leg-raise test (SLR) | Pre-intervention; Post-intervention (30 minutes after intervention); Follow up (4 week after last intervention)
  For the SLR test, a normal examination table is used. Participants lay supine and must be relaxed throughout the test. The tested limb is flexed by the examiner, with the knee fully extended and the foot in a relaxed position. The contralateral limb is secured by a second examiner, fully extended and in neutral rotation.
  The movement stops when the tester feels a strong resistance or when pelvic rotation is observed. The goniometer is placed over the greater trochanter, with 1 arm aligned with the lateral femoral condyle and the other aligned parallel to the table, in the direction of the midaxillary line.

SECONDARY OUTCOMES:
Change in Quadriceps Muscle Extensibility | Pre-intervention; Post-intervention (30 minutes after intervention); Follow up (4 week after last intervention)
  The assessor slowly bends the subject's knee so that the heel approximated the buttock. Attention is paid ensuring that there is no lumbar spine or pelvic movement or cramping of the hamstrings and that the thighs remained parallel. The subject is asked to report as soon as a first sensation of stretch is experienced in the quadriceps muscle. The closest distance from the relaxed buttock to the heel with the ankle passively plantar flexed, is measured with a goniometer. By holding the ankle and the weight of the lower leg, the assessor ensures that the quadriceps is itself not stretched in any way during this procedure as this could be interpreted as a treatment, rather than assessment.
Change in Frequency | Pre-intervention; Post-intervention (30 minutes after intervention); Follow up (4 week after last intervention)
  Frequency of muscle oscillations (Hz) is an indicator of the tone.This outcome measure is obtained by a device named MyotonPro. It is a non-invasive commercial device made to calculate myotonometrics properties of the muscle.
Change in Stiffness | Pre-intervention; Post-intervention (30 minutes after intervention); Follow up (4 week after last intervention)
  The muscle stiffness reflects muscle resistance to the force that changes its shape (Nm). This outcome measure is obtained by a device named MyotonPro. It is a non-invasive commercial device made to calculate myotonometrics properties of the muscle.
Change in Decrement (elasticity) | Pre-intervention; Post-intervention (30 minutes after intervention); Follow up (4 week after last intervention)
  Logarithmic decrement of the dampening of muscle oscillations is an indicator of the elasticity. This outcome measure is obtained by a device named MyotonPro. It is a non-invasive commercial device made to calculate myotonometrics properties of the muscle.
Change in Neural Measures | Pre-intervention; Post-intervention (30 minutes after intervention); Follow up (4 week after last intervention)
  To begin the test, patient must be seated with hands behind back to achieve a neutral spine. The first step is to have the patient slump forward at the thoracic and lumbar spine. If this position does not cause pain, patient must flex the neck by placing the chin on the chest and then extending one knee as much as possible.
  If extending the knee causes pain, patient must extend the neck into neutral. If the patient is still unable to extend the knee due to pain, the test is considered positive.
  If extending the knee does not cause pain, patient must do actively dorsiflexion of the ankle. If dorsiflexion causes pain, have the patient slightly flex the knee while still dorsiflexing. If the pain is reproduced, the test is considered positive.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Ortiz-Lucas, Principal Investigator — Universidad San Jorge
Locations (1):
- Universidad San Jorge, Villanueva de Gállego, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No